CLINICAL TRIAL: NCT03229850
Title: Dynamics of Insulin Absorption in Subclinical Lipohypertrophy Using the Euglycemic Clamp Technique
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was suspended due to current COVID 19 research curtailment
Sponsor: Graydon Meneilly (Other)
Responsible Party: Sponsor-Investigator, Graydon Meneilly, Professor, UBC Department of Medicine, University of British Columbia
Organization: University of British Columbia (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: H17-01270
Record Dates: First submitted 2017-06-26; First posted 2017-07-26 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Diabetes Mellitus; Lipohypertrophy
Keywords: Diabetes; Insulin; Lipohypertrophy; Euglycemic Clamp
MeSH Terms: conditions — Diabetes Mellitus; Insulin Resistance | interventions — Insulin Lispro

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: During one euglycemic clamp study, insulin lispro will be injected subcutaneously into an area of subclinical lipohypertrophy of the abdomen identified by ultrasound, during the other insulin lispro will be injected to an area with no subclinical lipohypertrophy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Subclinical Lipohypertrophy (Other): Insulin lispro will be injected in the abdomen into an area of subclinical lipohypertrophy.
  Interventions: Drug: Insulin lispro
- No Subclinical Lipohypertrophy (Other): Insulin lispro will be injected in the abdomen into an area where there is no subclinical lipohypertrophy.
  Interventions: Drug: Insulin lispro

INTERVENTIONS:
Drug: Insulin lispro — Insulin lispro will be injected into the abdomen into an area of subclinical lipohypertrophy or an area with no subclinical lipohypertrophy

SUMMARY:
This study will use the euglycemic clamp technique to evaluate insulin absorption when insulin is administered subcutaneously in an area of subclinical lipohypertrophy vs an area of normal tissue.

DETAILED DESCRIPTION:
The use of insulin to manage diabetes can cause changes to the skin at sites where insulin is administered. These changes may be felt as lumps under the skin. Insulin injected into these areas may not work as well leading to needing increasing doses of insulin to control blood glucose levels. Hypoglycemia can occur when insulin is injected into normal areas. Previous studies have found that these lipohypertrophic areas can be seen on ultrasound before they can be felt. The Investigators will be using the euglycemic clamp techique to evaluate insulin absorption to see whether tissue with lumps that cannot be felt but are seen on ultrasound affect how insulin is absorbed.

ELIGIBILITY:
Inclusion Criteria:

* Participated in Glycemic Variability study
* Type 2 Diabetes for at least 2 years
* Currently using insulin to manage diabetes
* Have used insulin to manage diabetes for at least 2 years
* Age 19 or older
* BMI < 30 kg/m2
* Confirmed areas of subclinical lipohypertrophic adipose tissue lesions via ultrasound

Exclusion Criteria:

* Taking other injectable medications (eg liraglutide/Victoza
* Taking systemic steroids (ie prednisone)
* Severe renal insufficiency (eGFR < 30 ml/min/1.73 m2
* Hypoglycemic unawareness
* Current pregnancy
* Not fluent in speaking and writing English (unless accompanied by a translator)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-04-22 (Actual)

PRIMARY OUTCOMES:
Insulin Levels | 2 months
  The euglycemic clamp technique will be used. Insulin levels will be analyzed by Eliza assay

CONTACTS AND LOCATIONS:
Overall Officials: Graydon Meneilly, MD, Principal Investigator — University of British Columbia
Locations (1):
- University of British Columbia - Gerontology Research Lab, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fujikura J, Fujimoto M, Yasue S, Noguchi M, Masuzaki H, Hosoda K, Tachibana T, Sugihara H, Nakao K. Insulin-induced lipohypertrophy: report of a case with histopathology. Endocr J. 2005 Oct;52(5):623-8. doi: 10.1507/endocrj.52.623. PMID 16284443
- [Background] Raile K, Noelle V, Landgraf R, Schwarz HP. Insulin antibodies are associated with lipoatrophy but also with lipohypertrophy in children and adolescents with type 1 diabetes. Exp Clin Endocrinol Diabetes. 2001;109(8):393-6. doi: 10.1055/s-2001-18991. PMID 11748486
- [Background] Schiazza L, Occella C, Bleidl D, Rampini E. Insulin lipohypertrophy. J Am Acad Dermatol. 1990 Jan;22(1):148-9. doi: 10.1016/s0190-9622(08)80037-0. No abstract available. PMID 2076114
- [Background] Vardar B, Kizilci S. Incidence of lipohypertrophy in diabetic patients and a study of influencing factors. Diabetes Res Clin Pract. 2007 Aug;77(2):231-6. doi: 10.1016/j.diabres.2006.12.023. Epub 2007 Feb 15. PMID 17303282
- [Background] Young RJ, Hannan WJ, Frier BM, Steel JM, Duncan LJ. Diabetic lipohypertrophy delays insulin absorption. Diabetes Care. 1984 Sep-Oct;7(5):479-80. doi: 10.2337/diacare.7.5.479. PMID 6389062
- [Background] Chowdhury TA, Escudier V. Poor glycaemic control caused by insulin induced lipohypertrophy. BMJ. 2003 Aug 16;327(7411):383-4. doi: 10.1136/bmj.327.7411.383. No abstract available. PMID 12919996
- [Background] Hauner H, Stockamp B, Haastert B. Prevalence of lipohypertrophy in insulin-treated diabetic patients and predisposing factors. Exp Clin Endocrinol Diabetes. 1996;104(2):106-10. doi: 10.1055/s-0029-1211431. PMID 8740933
- [Background] Blanco M, Hernandez MT, Strauss KW, Amaya M. Prevalence and risk factors of lipohypertrophy in insulin-injecting patients with diabetes. Diabetes Metab. 2013 Oct;39(5):445-53. doi: 10.1016/j.diabet.2013.05.006. Epub 2013 Jul 22. PMID 23886784
- [Background] Thow JC, Johnson AB, Marsden S, Taylor R, Home PD. Morphology of palpably abnormal injection sites and effects on absorption of isophane(NPH) insulin. Diabet Med. 1990 Nov;7(9):795-9. doi: 10.1111/j.1464-5491.1990.tb01494.x. PMID 2148131
- [Background] Overland J, Molyneaux L, Tewari S, Fatouros R, Melville P, Foote D, Wu T, Yue DK. Lipohypertrophy: does it matter in daily life? A study using a continuous glucose monitoring system. Diabetes Obes Metab. 2009 May;11(5):460-3. doi: 10.1111/j.1463-1326.2008.00972.x. Epub 2009 Feb 19. PMID 19236441
- [Background] Heinemann L, Weyer C, Rauhaus M, Heinrichs S, Heise T. Variability of the metabolic effect of soluble insulin and the rapid-acting insulin analog insulin aspart. Diabetes Care. 1998 Nov;21(11):1910-4. doi: 10.2337/diacare.21.11.1910. PMID 9802742
- [Background] Famulla S, Hovelmann U, Fischer A, Coester HV, Hermanski L, Kaltheuner M, Kaltheuner L, Heinemann L, Heise T, Hirsch L. Insulin Injection Into Lipohypertrophic Tissue: Blunted and More Variable Insulin Absorption and Action and Impaired Postprandial Glucose Control. Diabetes Care. 2016 Sep;39(9):1486-92. doi: 10.2337/dc16-0610. Epub 2016 Jul 13. PMID 27411698